CLINICAL TRIAL: NCT02674945
Title: Understanding and Improving Quality of Life Through a Wireless Activity Tracker: Observational Phase
Status: Terminated | Type: Observational
Why Stopped: Low enrollment, unable to power adequately
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1406M51644; #2014NTLS054 (Other: CPRC)
Record Dates: First submitted 2016-01-04; First posted 2016-02-05 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Brain Tumor
Keywords: fitbit; activity tracker; sleep; quality of life
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Wireless Activity tracker: Fitbit: Patients with brain tumor(s) will be give a wireless activity tracker (fitbit flex) to use during treatment. They will complete quality of life surveys and a sleep survey.
  Interventions: Device: Wireless Activity tracker: Fitbit

INTERVENTIONS:
Device: Wireless Activity tracker: Fitbit — Patients will wear a Fitbit flex

SUMMARY:
This project attempts to correlate wireless activity data with quality of life and sleep surveys in order to find a new method of monitoring patients during their treatment.

DETAILED DESCRIPTION:
This project proposes the investigation, validation, and use of a wireless activity tracker to better understand and improve the quality of life of patients suffering from brain tumors. The Fitbit flex wireless syncing activity tracker will be distributed to 75 patients, and the electronic infrastructure to automatically track patients will be created and adapted for the cohort. Surveys will routinely assess the ease-of-use and any problems arising. This heterogenous population of patients suffering from brain tumors will be tracked and compared through routine evaluation of their quality of life through well-established surveys, including the SF-36 and FACT-Br. The association between data recorded from the activity tracker and the QOL surveys will be quantified to validate the activity tracking data as a surrogate measure of part, if not all, of QOL as well as sleep.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with primary or metastatic brain tumor
* able to wear wireless activity tracker
* able to complete QOL and sleep surveys every 3 months

Exclusion Criteria:

* unable to provide consent
* age < 18
* lack of use of the wireless activity tracker for more than 2 consecutive months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consentable patients suffering from a single or multiple primary or metastatic brain tumors
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Activity measured in steps | 1 year delineated by minute

SECONDARY OUTCOMES:
Sleep | per night over 1 year
  wireless activity will attempt to monitor sleep cycles when the device is worn
Quality of Life - SF-36 | months 0, 3, 6, 9, and 12
  SF-36
Quality of Life - Fact- Br | months 0, 3, 6, 9, and 12
  Fact-Br

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared. De-identified group data will be made available